CLINICAL TRIAL: NCT03999814
Title: A Retrospective Review of the Natural History of Infantile Neuroaxonal Dystrophy
Brief Title: Natural History of Infantile Neuroaxonal Dystrophy
Status: Completed | Type: Observational
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RT-INAD-NH001
Record Dates: First submitted 2019-04-25; First posted 2019-06-27 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2019-06

CONDITIONS: Infantile Neuroaxonal Dystrophy; INAD
Keywords: Infantile Neuroaxonal Dystrophy; INAD; PLA2G6
MeSH Terms: conditions — Neuroaxonal Dystrophies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective and cross-sectional review of the natural history of INAD.

DETAILED DESCRIPTION:
After obtaining informed consent, the study participants' relevant medical records will be collected and reviewed. If needed, a telephone or video conference will be scheduled with the patient's family to confirm and clarify information in the medical record. Deceased patients may be eligible for inclusion the retrospective registry if medical records are sufficient and indicate eligibility. Data will be pooled and presented in aggregate, without identification of individual subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 months to 10 years of age
* Medical history consistent with the symptoms of classic INAD (onset of symptoms between the ages of 6 months and 3 years)
* Homozygous for PLA2G6 deficiency (variant alleles may be mixed heterozygotes)
* Signed informed consent form (ICF) prior to entry into the registry

Exclusion Criteria:

* Diagnosis of atypical NAD (ANAD)
* Unwilling or unable to allow medical record review

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Living or deceased males or females with a diagnosis of classic INAD between the ages of 18 months and 10 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
To describe the natural history of infantile neuroaxonal dystrophy (INAD). | Birth to time of enrollment.
  Overall analysis

SECONDARY OUTCOMES:
To look for trends in disease progression of INAD that may be helpful in planning future interventional trials in INAD. | Birth to time of enrollment.
  Overall analysis
Evaluating and potentially validating a Assessment of Severity by Parent or Caregiver questionnaire. | At time of enrollment.
  In the questionnaire parents/caregivers are asked to score the child on a scale of 1 to 4 based on how often the child can perform 33 various activities of daily living. The individual scores are then added up to form a composite score of disease severity, with lower scores indicating higher severity and higher score indicating less disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milner, MD, Principal Investigator — Biojiva LLC
Locations (1):
- Sarah Endemann, Los Altos, California, United States

IPD SHARING:
Plan to Share IPD: No